CLINICAL TRIAL: NCT01741545
Title: A Phase 3 Study Evaluating the Safety and Efficacy of Lambda/Ribavirin/Daclatasvir in Subjects With Chronic HCV Infection and Underlying Hemophilia Who Are Treatment Naïve or Are Prior Relapsers to Peginterferon Alfa-2a/Ribavirin
Brief Title: Safety and Efficacy Study in Subjects With Chronic HCV and Underlying Hemophilia
Acronym: MAGNITUDE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI452-030; 2012-003463-22 (EudraCT Number)
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon lambda-1a; Ribavirin; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A: Genotype-2,-3 (Lambda/RBV/DCV) (Experimental): Lambda 180 μg solution for subcutaneous (SC) injection, once weekly for 12 weeks
  Ribavirin (RBV) 200 mg tablet by mouth (oral), twice daily for 12 weeks
  Daclatasvir (DCV) 60mg tablet by mouth (oral), once daily for 12 weeks
  Interventions: Biological: Pegylated-Interferon-lambda; Drug: Ribavirin; Drug: Daclatasvir
- Cohort B: Genotype-1b,-4 (Lambda/RBV/DCV) (Experimental): Lambda 180 μg solution for subcutaneous (SC) injection, once weekly for 24 weeks
  Ribavirin (RBV) 200 mg tablet by mouth (oral), twice daily for 24 weeks
  Daclatasvir (DCV) 60mg tablet by mouth (oral), once daily for 12 weeks
  Interventions: Biological: Pegylated-Interferon-lambda; Drug: Ribavirin; Drug: Daclatasvir

INTERVENTIONS:
Biological: Pegylated-Interferon-lambda
  Other Names: pegIFNλ; BMS-914143
Drug: Ribavirin
Drug: Daclatasvir
  Other Names: BMS-790052

SUMMARY:
The primary objective for this study is to evaluate the proportion of subjects who achieve SVR12 (HCV RNA < LLOQ (target not detected) at post-treatment follow-up Week 12 in subjects with Genotype(GT)-1b, -4 and GT-2, -3

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Severe hemophilia (defined as < 1% factor activity level)
* Infection with the hepatitis C virus (HCV) with underlying hemophilia
* Males 18 years of age and above
* Have not been previously treated with an interferon

Exclusion Criteria:

* Not infected with the hepatitis B virus (HBV) or human immunodeficiency virus (HIV)
* Chronic liver disease caused by any disease other than chronic HCV infection
* Presence of Bethesda inhibitor
* Current evidence of or history of portal hypertension

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2013-03-31 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2015-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (30):
- United States (4):
  - Stanford Boswell Clinic, Palo Alto, California
  - Rush University Medical Center, Chicago, Illinois
  - Hospital Of The University Of Pennsylvania, Philadelphia, Pennsylvania
  - Clinical Research Centers Of America, Murray, Utah
- Australia (5):
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Herston, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Melbourne, Victoria
  - Local Institution, Herston
- France (5):
  - Local Institution, Grenoble
  - Local Institution, Lyon
  - Local Institution, Montpellier
  - Local Institution, Paris
  - Local Institution, Vandœuvre-lès-Nancy
- Italy (4):
  - Local Institution, Florence
  - Local Institution, Milan
  - Local Institution, Roma
  - Local Institution, Torino
- Netherlands (4):
  - Local Institution, Amsterdam
  - Local Institution, Nijmegen
  - Local Institution, Rotterdam
  - Local Institution, Utrecht
- Romania (3):
  - Local Institution, Bucharest
  - Local Institution, Constanța
  - Local Institution, Iași
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- Spain (3):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Seville

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 71 participants were enrolled, of which 51 subjects were randomized and treated.
Groups:
- Cohort A: Participants with hepatitis C virus (HCV) genotype (GT)-2 or GT-3 infection (Cohort A) were treated with peginterferon lambda-1a (pegIFNλ-1a referred to as Lambda)/Ribavirin (RBV)/Daclatasvir (DCV). Participants were administered daclatasvir 60 mg orally, once daily; peginterferon lambda-1a 180 microgram subcutaneous injection, once weekly and ribavirin tablets, orally, twice daily (a total 800 mg per day) for 12 weeks treatment, 12 weeks and a maximum of 12 weeks, respectively (treatment period= 12 Weeks). Participants were followed up for 24 weeks after administration of last treatment (follow-up period= 24 Weeks).
- Cohort B: Participants with HCV GT-1b or GT-4 infection (Cohort B) were treated with Lambda/Ribavirin/Daclatasvir. Participants were administered daclatasvir 60 mg orally, once daily, peginterferon lambda-1a 180 microgram subcutaneous injection, once weekly and ribavirin tablets, twice daily, orally, based on weight (participants weighing <75 kg = 1000 mg and participants weighing >=75 kg = 1200 mg per day) for 12 weeks treatment, 24 weeks and a maximum of 24 weeks, respectively (treatment period= 24 Weeks). Participants were followed up for 24 weeks after administration of last treatment (follow-up period= 24 Weeks).
Period: Treatment Period
Arm/Group | Cohort A | Cohort B
Started | 12 | 39
Completed | 11 | 35
Not Completed | 1 | 4
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse event, non-fatal | 1 | 3
Period: Follow-up Period (24 Weeks)
Arm/Group | Cohort A | Cohort B
Started | 12 (1 participant re-joined Cohort A in follow-up period.) | 39 (4 participants re-joined Cohort B in follow-up period.)
Completed | 11 | 37
Not Completed | 1 | 2
Not completed — Other than specified | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: All treated participants.
Groups:
- Cohort A: Participants with HCV GT-2 or GT-3 infection (Cohort A) were treated with Lambda/Ribavirin/Daclatasvir. Participants were administered daclatasvir 60 mg orally, once daily; peginterferon lambda-1a 180 microgram subcutaneous injection, once weekly and ribavirin tablets, orally, twice daily (a total 800 mg per day) for 12 weeks treatment, 12 weeks and a maximum of 12 weeks, respectively (treatment period= 12 Weeks). Participants were followed up for 24 weeks after administration of last treatment (follow-up period= 24 Weeks).
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 12 | 39 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 38 | 50
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (9.94) | 45.2 (12.04) | 44.6 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 39 | 51
HCV Genotype [Count of Participants; unit: Participants]
  Genotype 1A | 0 | 0 | 0
  Genotype 1B | 0 | 39 | 39
  Genotype 2 | 2 | 0 | 2
  Genotype 3 | 10 | 0 | 10
  Genotype 4 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Sustained Virologic Response (SVR12) at Follow-Up Week 12
Description: SVR12 was defined as HCV ribonucleic acid (RNA) less than the lower limit of quantitation, target detected or target not detected at follow-up Week 12.
Time Frame: Follow-up Week 12
Population: The analysis was performed in modified intent to treat (mITT) population defined as participants meeting the response criteria over all treated participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 39
Percentage of participants | 91.7 [61.5 to 99.8] | 89.7 [75.8 to 97.1]

2. Secondary Outcome: Percentage of Participants With Rapid Virologic Response (RVR)
Description: RVR was defined as HCV RNA less than the lower limit of quantitation, target not detected at Week 4.
Time Frame: Treatment Week 4
Population: mITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 39
Percentage of participants | 91.7 [61.5 to 99.8] | 76.9 [60.7 to 88.9]

3. Secondary Outcome: Percentage of Participants With Complete Early Virologic Response (cEVR)
Description: cEVR was defined as HCV RNA less than the lower limit of quantitation, target not detected at Week 12.
Time Frame: Treatment Week 12
Population: mITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 39
Percentage of participants | 91.7 [61.5 to 99.8] | 92.3 [79.1 to 98.4]

4. Secondary Outcome: Percentage of Participants With End of the Treatment Response (EOTR)
Description: EOTR was defined as HCV RNA less than the lower limit of quantitation, target not detected at end of treatment.
Time Frame: End of the treatment (Week 12 for Cohort A, Week 24 for Cohort B)
Population: mITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 39
Percentage of participants | 100 [73.5 to 100] | 100 [91 to 100]

5. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at Follow-Up Week 24 (SVR24)
Description: SVR24 was defined as HCV RNA less than the lower limit of quantitation, target detected or target not detected at follow-up week 24.
Time Frame: Follow-up Week 24
Population: mITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 39
Percentage of participants | 66.7 [34.9 to 90.1] | 30.8 [17 to 47.6]

6. Secondary Outcome: Percentage of Participants With Treatment-Emergent Cytopenic Abnormalities On-Treatment
Description: Cytopenic abnormalities were defined as anemia: Hemoglobin (Hb) <10 g/dL, and/or neutropenia: absolute neutrophils and bands (ANC) <750 mm^3, and/or thrombocytopenia: platelets <50,000 mm^3.
Time Frame: After day 1 to end of treatment (Up to 85 Days for Cohort A, Up to 168 Days for Cohort B)
Population: mITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 39
Percentage of participants | 0 [0 to 26.5] | 0 [0 to 9]

7. Secondary Outcome: Percentage of Participants With Flu-Like Symptoms and Musculoskeletal Symptoms On-Treatment
Description: Flu-like symptoms were defined as pyrexia or chills or pain. Musculoskeletal symptoms were defined as arthralgia or myalgia or back pain.
Time Frame: After day 1 to end of treatment (Up to 85 Days for Cohort A, Up to 168 Days for Cohort B)
Population: mITT population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 39
Percentage of participants
  Flu-like symptoms | 8.3 [0.2 to 38.5] | 12.8 [4.3 to 27.4]
  Musculoskeletal symptoms | 0 [0 to 26.5] | 15.4 [5.9 to 30.5]

8. Secondary Outcome: Percentage of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), AEs Leading to Discontinuation, Dose Reductions, And Death
Description: AE=any new untoward medical event or worsening of a preexisting medical condition that does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event. Treatment-related SAE=possibly, probably, or certainly related to study drug.
Time Frame: From Day 1 to end of follow-up (maximum of 60 weeks for Cohort A and 72 weeks for Cohort B)
Population: All treated participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 39
Percentage of participants
  AEs on treatment | 10 | 38
  SAEs | 0 | 4
  Death | 0 | 0
  AE leading to discontinuation | 1 | 3
  Dose reduction - Lambda | 0 | 1
  Dose reduction - RBV | 0 | 2

9. Secondary Outcome: Number of Participants With Treatment Emergent Grade 3 to 4 Laboratory Abnormalities
Description: Laboratory abnormalities were determined and graded using the Division of acquired immunodeficiency syndrome (AIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, version 1.0. International Normalized Ratio (INR): >2.0*Upper limit of normal (ULN); Alanine aminotransferase (ALT) : >5*ULN; Aspartate aminotransferase (AST): >5*ULN; Prothrombin Time (PT): >1.50*ULN; Bilirubin (Total): >2.5*ULN; Triglycerides (fasting): >750 mg/dL.
Time Frame: After day 1 to to end of treatment (Up to 85 Days for Cohort A, Up to 168 Days for Cohort B)
Population: All treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 12 | 39
Participants
  INR | 0 | 1
  ALT | 2 | 1
  AST | 0 | 2
  PT | 0 | 1
  Bilirubin | 2 | 7
  Triglycerides | 0 | 1

ADVERSE EVENTS:
Time Frame: From Day 1 to end of follow-up (maximum of 60 weeks for Cohort A and 72 weeks for Cohort B)
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/12 | 4/39
Other Adverse Events (participants affected / at risk) | 10/12 | 36/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=12) | Cohort B (N=39)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=12) | Cohort B (N=39)
Haematoma (Vascular disorders) | 0 (0) | 3 (3)
Haemorrhage (Vascular disorders) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 12 (12)
Fatigue (General disorders) | 3 (3) | 9 (9)
Pyrexia (General disorders) | 1 (1) | 5 (5)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 13 (13)
Sleep disorder (Psychiatric disorders) | 1 (1) | 5 (5)
Affect lability (Psychiatric disorders) | 0 (0) | 2 (2)
Anger (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Irritability (Psychiatric disorders) | 2 (2) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 2 (2)
Weight decreased (Investigations) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 1 (1)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 7 (7)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Disturbance in attention (Nervous system disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chromaturia (Renal and urinary disorders) | 2 (2) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (7)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submitting for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.